CLINICAL TRIAL: NCT01511302
Title: A Phase I, Single-Blinded, Randomized Study of Nebulized RNS60 in Combination With Budesonide in Adult Subjects With Mild to Moderate Asthma
Brief Title: Study of Inhaled RNS60 in Combination With Budesonide to Treat Mild to Moderate Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01.1.1.H2
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — RNS60; Saline Solution; Budesonide

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- RNS60-BD 0.25 (Experimental): RNS60 in combination with Budesonide 0.25mg/2ml concentration
  Interventions: Drug: RNS60; Drug: Budesonide
- RNS60-BD 0.5 (Experimental): RNS60 in combination with Budesonide 0.5mg/2ml concentration
  Interventions: Drug: RNS60; Drug: Budesonide
- NS-BD 0.5 (Placebo Comparator): Normal Saline control (NS) in combination with Budesonide 0.5mg/2ml concentration
  Interventions: Drug: Normal Saline; Drug: Budesonide

INTERVENTIONS:
Drug: RNS60 — RNS60, 2ml, nebulized twice daily.
  Arms: RNS60-BD 0.25; RNS60-BD 0.5
Drug: Normal Saline — Normal Saline placebo, 2 ml, nebulized twice daily.
  Arms: NS-BD 0.5
Drug: Budesonide — Budesonide, in either 0.25 mg or 0.5 mg per 2 ml concentration in liquid suspension, nebulized once per day in combination with RNS60 or NS.

SUMMARY:
The purpose of this study is to determine whether RNS60, in combination with budesonide, is safe in mild to moderate asthmatics when taken by nebulization over a 28-day period, compared to a 28-day control period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female non-smokers, aged between 18 and 65 years.
* Clinical diagnosis of mild to moderate asthma meeting NHLBI 2007 guidelines as outlined in Appendix A.
* Subjects who have a currently prescribed inhaled corticosteroid medication to treat asthma, alone or in combination with other medications, with usage of 1 month (≥ 95% compliance) or more on the inhaled corticosteroid treatment.
* Normal 12-lead ECG at Screening.
* Normal single view chest x-ray at Screening.
* Men and women of reproductive potential who commit to use adequate contraception during the study and for 1 month following the last day of treatment (Day 57).
* Women of childbearing potential who have a negative pregnancy test (serum HCG) at the time of study entry, and again on Day 22.
* Subjects, or their legal guardians, must be capable of understanding the purpose and risks of the study and provide written, voluntary, informed consent.

Exclusion Criteria:

* Chronic or acute disease that might interfere with the evaluation of RNS60.
* Pregnancy, intent to become pregnant, or breastfeeding.
* Current or prior malignancies (excluding non-melanoma skin carcinoma or in situ carcinoma of the cervix that has been adequately treated).
* Positive viral serology test for Human Immunodeficiency Virus (HIV-1), HBsAG and Hepatitis C antibody.
* Positive urine drug screen (UDS) for drugs of abuse including alcohol and cotinine at the time of study entry and again on Day 22.
* Infections that require intravenous antibiotic therapy.
* Significant organ dysfunction, including cardiac, renal, liver, central nervous system, pulmonary, vascular, gastrointestinal, endocrine, or metabolic (e.g., creatinine ≥ 1.6 mg/dL; ALT or AST ≥ 1.5x the upper limit of normal), history of myocardial infarction, congestive heart failure, or arrhythmias within 6 months prior to study entry.
* Treatment with a humanized or chimeric antibody therapy within 4 weeks prior to study entry.
* Treatment with any investigational drugs, therapies, or medical devices within 4 weeks prior to study entry.
* Any use of antidepressants or other psychiatric medicine within 4 weeks prior to study entry and/or during the study treatment period.
* Use of any over-the-counter asthma treatments, including Primatene Mist, during the 8-week active study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Forced expiratory volume in 1 second (FEV1) | Baseline to 56 days
  Evidence that RNS60 in combination with budesonide does not cause bronchoconstriction, as measured by FEV1 scores.

SECONDARY OUTCOMES:
Change in peak expiratory flow | Baseline to 56 days
  Evidence that RNS60 in combination with budesonide does not cause bronchoconstriction, as measured by daily peak expiratory flow values.
Change in quality of life | 56 days
  Evidence that RNS60 in combination with budesonide does not reduce patient's quality of life, as measured by weekly QOL questionnaire over 28 days.
Change in rescue inhaler usage | 56 days
  Evidence that RNS60 in combination with budesonide does not increase rescue inhaler usage, as measured by patient diary.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - West Coast Clinical Trials, Costa Mesa, California
  - California Allergy and Asthma, Los Angeles, California
  - Axis Clinical Trials, Los Angeles, California
  - Integrated Research Group, Riverside, California